CLINICAL TRIAL: NCT02050074
Title: The Role of Metformin and Colesevelam in Human GLP-1 Secretion
Acronym: ColMetInc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hansen, Dr., University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-1-2013-010
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Colesevelam (Experimental)
  Interventions: Drug: Colesevelam
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Placebo (Experimental)
  Interventions: Other: Placebo
- Colesevelam + exendin (9-39) (Experimental)
  Interventions: Drug: Colesevelam
- Metformin + exendin (9-39) (Experimental)
  Interventions: Drug: Metformin
- Placebo + + exendin (9-39) (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Colesevelam
  Arms: Colesevelam; Colesevelam + exendin (9-39)
Drug: Metformin
  Arms: Metformin; Metformin + exendin (9-39)
Other: Placebo
  Arms: Placebo; Placebo + + exendin (9-39)

SUMMARY:
Our primary hypothesis is that bile acid sequestrant colesevelam and the antidiabetic drug metformin potentiates the secretion of the gut hormone glucagon-like peptide 1 (GLP-1).

ELIGIBILITY:
Inclusion Criteria:

* Normal hemoglobin
* BMI > 23kg/m2
* HbA1c <9 %
* Informed concent

Exclusion Criteria:

* Liver disease ( aspartate aminotransferase/alanine aminotransferase >2 × reference value)
* Chronic intestinal disease
* History of liver and / or gallbladder disease
* Nephropathy (se-creatinine >110 µM and / or albuminuria)
* Insulin or GLP-1-based antidiabetic treatment
* History of cholecystectomy or surgical resection of bowel segment
* BMI <23kg/m2 or BMI >35 kg/m2
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in the gut hormone glucagon-like peptide 1 (GLP-1) | 0-240 min

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Division, Department of Medicine, Gentofte Hospital, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Derived] Bahne E, Sun EWL, Young RL, Hansen M, Sonne DP, Hansen JS, Rohde U, Liou AP, Jackson ML, de Fontgalland D, Rabbitt P, Hollington P, Sposato L, Due S, Wattchow DA, Rehfeld JF, Holst JJ, Keating DJ, Vilsboll T, Knop FK. Metformin-induced glucagon-like peptide-1 secretion contributes to the actions of metformin in type 2 diabetes. JCI Insight. 2018 Dec 6;3(23):e93936. doi: 10.1172/jci.insight.93936. PMID 30518693